CLINICAL TRIAL: NCT04063332
Title: Functionality of Endogenous Biological Clock in Sepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Athens (Other)
Collaborators: Hellenic Sepsis Study Group (Other)
Responsible Party: Principal Investigator, Evangelos J. Giamarellos-Bourboulis, M.D., MD, PhD, Professor of Internal Medicine ,President-Elect: European Shock Society, Co-ordinator: Hellenic Sepsis Study Group, University of Athens
Other Study IDs: CLOCK
Record Dates: First submitted 2019-08-13; First posted 2019-08-21 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Circadian Rhythm Disorders; Sepsis
Keywords: circadian; sepsis; clock; melatonin
MeSH Terms: conditions — Chronobiology Disorders; Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for mRNA analysis and hormones' measurements
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- GROUP A: Absolutely healthy individuals without any comorbidities, working at the same environment with the rest of groups (doctors are excluded as belong to one of the special categories) patients with sepsis as defined by the Sepsis-3 classification criteria3
- GROUP B: Control patients without sepsis or infection and with the same exactly comorbidities (ideally ≤2 suffering organ systems) , i.e. identical Charlson score, identical mental status and age difference ≤ 5 years with group A
- GROUP C: Patients with sepsis as defined by the Sepsis-3 classification criteria3

SUMMARY:
The aim of the current study is to demonstrate dysregulation of immune system΄s circadian rhythms as a consequence of sepsis, as well as marked malfunction of the central circadian clock in comparison with patients without sepsis , the presence of which burdens independently the final outcome and , hence, need to be addressed.

DETAILED DESCRIPTION:
Sepsis is number one cause of death within the critically ill patients ,with mortality that reaches a rate of 70%,while in case of the establishment of septic shock and multi organ failure it can rise up to 80%.Septic shock is the most common cause of death in the ICUs. It has been estimated that 25% of the total of septic patients will develop severe sepsis (sepsis and organ failure), while septic shock (sepsis and cardiovascular failure).

In order to call a biological rhythm circadian, the following 3 criteria must be satisfied:

1. Insistence on stable conditions, with endogenous period of about 24 hours.
2. Independence of ambient temperature, so that almost always progresses at the same rate (same frequency), independent of temperature.
3. This endogenous rhythm, of approximately 24 hours, can be synchronized in exactly 24 hours, influenced by environmental factors, such as light/dark cycles, social interactions, etc.

Many organic systems follow a circadian pattern, among others the immune system,on the grounds that peripheral blood lymphocytes own all the forementioned genes, whose coordinated expression with that particular periodicity results in the generation of maximum (peak) and minimum (nadir) of the number of circulating cells, their activity, the production and secretion of cytokines etc.This endogenous attitude is lost in case of sepsis, due to few or absent stimuli deriving from the central clock. As a result, an additional compounding factor comes up in the immune system ,which fails to fight the infectious agent and that inefficient immune response aggravates the circadian desynchronization , creating a vicious circle.

The direct evaluation of circadian rhythms' entails the examination of suprachiasmatic neurons' functionality, through biopsies from the examined patients ,which constitutes an ethically questionable ,practically expensive, time-consuming and quite demanding procedure. Thus, the estimation of actual circadian profile will take place indirectly, driven by a series of biomarkers, indicative of the functional status of the ''central biological clock'' found at the suprachiasmatic nucleus of CNS (melatonin, cortisol, core body temperature),as well as the ''peripheral clock'' placed at the immune system cells (Clock/ Bmal1 , Per/Cry genes' expression).

The purpose of this prospective, observational, case-control study is to investigate the discrepancy in levels of circadian biomarkers in patients suffering from sepsis in comparison with those coming from other ,non-septic patients in the same environment as well as deviation from healthy controls' values, and secondarily to assess the effect of septic syndrome in later development of endogenous clock that regulates daily life with regard to the quality of life that follows recovery.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥18 years)
* Written informed consent
* Male or female gender
* Οne of the following cases:

  * Healthy controls without comorbidities OR
  * Patients without sepsis or infection , with identical Charlson Comorbidity Index and same mental status with the septic patients OR
  * Patients with sepsis

Exclusion Criteria:

* Failure to obtain written informed consent
* Age <18 years
* Pregnancy or breastfeeding
* Solid tumor or hematologic malignancy
* Asthma
* Neurodegenerative disease
* Traumatic brain injury
* Confirmed depression
* Autoimmune disorders
* Special categories following unfixed or varying routine schedules (e.g. travels overseas or even short distances, if frequent/jet lag/on-call duties/nightshifts with regard to doctors,security guards,singers)
* Per os or iv corticosteroids daily intake of dose at least
* Corticosteroid oral or intravenous intake of at least 0.4 mg/kg of equivalent prednisone daily over the last 15 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * GROUP A: absolutely healthy individuals without any comorbidities, working at the same environment with the rest of groups (doctors are excluded as belong to one of the special categories) patients with sepsis as defined by the Sepsis-3 classification criteria3
  * GROUP Β: control patients without sepsis or infection and with the same exactly comorbidities (ideally ≤2 suffering organ systems) , i.e. identical Charlson score, identical mental status and age difference ≤ 5 years with group A
  * GROUP C: patients with sepsis as defined by the Sepsis-3 classification criteria3
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-06-03 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
The substantial discrepancy in the values of melatonin, cortisol and core body temperature (central CLOCK circadian markers) between septic and non-septic patients. | 7 days
  Different values in melatonin,cortisol, core body temperature .
The substantial discrepancy in the circadian rhythms' genes expression levels (peripheral clock markers) between septic and non-septic patients ,within their peripheral blood leucocytes . | 7 days
  Different mRNA levels of clock, bmal1, per, cry genes within peripheral blood leucocytes.
The difference in the extent of deviation from normal, with regard to the values of melatonin-cortisol-core body temperature (circadian triad) between septic and non-septic patients. | 7 days
  Extent of abnormality in the values of melatonin,cortisol and core body temperature .
The difference in the extent of deviation from normal, with regard to the levels of circadian rhythms' genes expression (immune system's clock) between septic and non-septic patients ,within their peripheral blood leucocytes . | 7 days
  Extent of abnormality in the mRNA levels of clock, bmal1, per, cry genes within peripheral blood leucocytes.

SECONDARY OUTCOMES:
Mortality rate at 28 days. | 28 days
  Differences in early (28-day) all-cause mortality rate between septic and matched non-septic patients .
Mortality rate at 90 days. | 90 days
  Differences in middle term (90-day) all-cause mortality rate between septic and matched non-septic patients.
Munich ChronoType Questionnaire results ,including Mid-sleep, Sleep Duration on both work and free days (MSw, MSf, MSfsc, SLDw, SLDf, SLDØ, chronotype). | 30 days
  Rate of circadian physiology restoration, concerning the discharged subgroup which is recovering from sepsis, with regard to daily routine and quality of life.
Pittsburgh Sleep Quality Index (Global PSQI Score). | 30 days
  Sum (range 0 to 21) of seven components,each scored 0 (no difficulty) to 3 (severe difficulty).These entail Subjective sleep quality, Sleep latency, duration, efficiency and disturbance, in addition to Use of sleep medication and Daytime dysfunction.
Munich ChronoType Questionnaire results ,including Mid-sleep, Sleep Duration on both work and free days (MSw, MSf, MSfsc, SLDw, SLDf, SLDØ, chronotype). | 60 days
  Rate of circadian physiology restoration ,concerning the discharged subgroup which is recovering from sepsis, with regard to daily routine and quality of life.
Pittsburgh Sleep Quality Index (Global PSQI Score). | 60 days
  Sum (range 0 to 21) of seven components,each scored 0 (no difficulty) to 3 (severe difficulty).These entail Subjective sleep quality, Sleep latency, duration, efficiency and disturbance, in addition to Use of sleep medication and Daytime dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos J Giamarellos-Bourboulis, MD, PhD, Principal Investigator — University of Athens
Locations (2):
- Greece (2):
  - 2nd Department of Intensive Care Medicine, Attikon University Hospital, Athens, Attica
  - 4th Department of Internal Medicine, Attikon University Hospital, Athens, Attica